CLINICAL TRIAL: NCT00071929
Title: Phase II Evaluation of Oxaliplatin in the Treatment of Recurrent or Persistent Endometrial Carcinoma
Brief Title: Oxaliplatin in Treating Patients With Persistent or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068235; GOG-0129K
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2004-09

CONDITIONS: Endometrial Cancer
Keywords: recurrent endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of oxaliplatin in treating patients who have persistent or recurrent endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of oxaliplatin in terms of response rate in patients with persistent or recurrent endometrial carcinoma that is refractory to curative or established therapy.
* Determine the nature and degree of toxicity of this treatment regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oxaliplatin IV over 2 hours on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: Approximately 19-51 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed endometrial carcinoma that is refractory to curative therapy or established treatment

  * Clinically and/or histologically confirmed persistent or recurrent disease
* Measurable disease by physical examination or medical imaging

  * Sonography allowed if lesions are clearly defined on initial examination and bidimensionally measurable
  * Ascites or pleural effusions not considered measurable
* Must have received 1 prior cytotoxic therapy regimen

  * May include high-dose therapy, consolidation, or extended therapy after surgical or nonsurgical assessment
  * 1 additional noncytotoxic regimen allowed

    * Biologic or cytostatic agents include, but are not limited to:

      * Monoclonal antibodies
      * Cytokines
      * Small-molecule inhibitors of signal transduction
* Ineligible for a higher priority GOG protocol
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* GOG 0-2 if received 1 prior therapy regimen
* GOG 0-1 if received 2 prior therapy regimens

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* No symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia

Neurologic

* No sensory or motor neuropathy greater than grade 1
* No residual neuropathy attributed to prior chemotherapy or other chronic conditions (e.g., diabetes, venous stasis, or carpal tunnel syndrome)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergy to platinum compounds or antiemetics
* No active infection requiring antibiotics
* No other uncontrolled illness
* No other invasive malignancies within the past 5 years except nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 14 days since prior pegfilgrastim
* At least 24 hours since other prior growth factors
* At least 3 weeks since prior biologic or immunologic therapy
* No concurrent growth factors during first course of study therapy

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy and recovered
* No more than 1 prior cytotoxic chemotherapy regimen, either single or combination cytotoxic drug therapy
* No prior oxaliplatin

Endocrine therapy

* At least 1 week since prior hormonal therapy directed at tumor
* Concurrent hormone replacement therapy allowed

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered

Surgery

* Recovered from any recent surgery

Other

* At least 3 weeks since prior therapy for endometrial cancer
* No other concurrent investigational agents
* No prior anticancer therapy that would preclude study participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-11; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula M. Fracasso, MD, PhD, Study Chair — Washington University Siteman Cancer Center
Locations (38):
- United States (38):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - New Britain General Hospital, New Britain, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Southeast Gynecologic Oncology Associates, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas

REFERENCES:
- [Result] Fracasso PM, Blessing JA, Molpus KL, Adler LM, Sorosky JI, Rose PG. Phase II study of oxaliplatin as second-line chemotherapy in endometrial carcinoma: a Gynecologic Oncology Group study. Gynecol Oncol. 2006 Nov;103(2):523-6. doi: 10.1016/j.ygyno.2006.03.043. Epub 2006 May 19. PMID 16712905